CLINICAL TRIAL: NCT03740737
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Groups, Multicenter Trial Investigating the Efficacy and Safety of FE 999049 in Controlled Ovarian Stimulation in Women Aged 18-34 Years Undergoing Assisted Reproductive Technology
Brief Title: Recombinant FSH Investigation in the Treatment of Infertility With Assisted Reproductive Technology (ART) (RITA-1)
Acronym: RITA-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000001
Record Dates: First submitted 2018-10-24; First posted 2018-11-14 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — follitropin delta; FE 999049

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FE 999049 (Follitropin Delta) (Experimental)
  Interventions: Drug: Follitropin delta
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Follitropin delta — FE 999049 was administered as single daily subcutaneous injections in the abdomen at a starting dose of 12 µg daily that was fixed for the first four stimulation days. Based on ovarian response, the dose could be adjusted by 3 µg, with dose increases implemented not more frequently than once every 2 days and dose decreases implemented per investigator's judgement. The minimum daily dose was 6 µg, and the maximum daily dose was 24 µg.
  Participants could be treated for a maximum of 20 days. Coasting, use of dopamine agonist or any other drug to prevent early ovarian hyperstimulation syndrome (OHSS) with the exception of gonadotropin-releasing hormone (GnRH) agonist for triggering of final follicular maturation, was not allowed.
  Other Names: FE 999049; Rekovelle
  Arms: FE 999049 (Follitropin Delta)
Other: Placebo — Placebo was administered as single daily subcutaneous injection dialed to the same value (dose) as FE 999049.
  Participants could be treated for a maximum of 20 days. Coasting, use of dopamine agonist or any other drug to prevent early OHSS with the exception of GnRH agonist for triggering of final follicular maturation, was not allowed.
  Arms: Placebo

SUMMARY:
This trial investigates the effects of FE 999049 compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Documents signed prior to any trial-related procedure.
* In good physical and mental health in the judgement of the investigator.
* Pre-menopausal females between the ages of 18 and 34 years. The participants must be at least 18 years (including the 18th birthday) when they sign the informed consent and no more than 34 years (up to the day before the 35th birthday) at the time of randomization.
* Body mass index (BMI) between 17.5 and 38.0 kg/m2 (both inclusive) at screening.
* Infertile women diagnosed with tubal infertility, unexplained infertility, endometriosis stage I/II or with partners diagnosed with male factor infertility, eligible for in vitro fertilization (IVF) and/or intracytoplasmic sperm injection (ICSI) using fresh or frozen ejaculated sperm from male partner or sperm donor.
* Documented history of infertility for at least 12 months before randomization (not applicable in case of tubal or severe male factor infertility, or when the use of donor sperm is indicated).
* Regular menstrual cycles of 24-35 days (both inclusive).
* Hysterosalpingography, hysteroscopy or saline infusion sonography, documenting a uterus consistent with expected normal function (e.g. no evidence of clinically interfering uterine fibroids defined as submucous fibroids of any size or intramural fibroids larger than 3 cm in diameter, no polyps and no congenital structural abnormalities which are associated with a reduced chance of pregnancy) at screening or within 1 year prior to screening.
* Transvaginal ultrasound documenting presence and adequate visualization of both ovaries, without evidence of significant abnormality (e.g. enlarged ovaries which would contraindicate the use of gonadotropins) and normal adnexa (e.g. no hydrosalpinx) at screening. Both ovaries must be accessible for oocyte retrieval.
* Early follicular phase (cycle day 2-4) serum levels of FSH between 1 and 15 IU/L (results obtained within 3 months prior to randomization).
* Negative serum Hepatitis B Surface Antigen (HBsAg), Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV) antibody tests at screening or within 6 months prior to screening.
* Willing to accept single blastocyst transfer in the fresh cycle and in the cryopreserved cycles initiated within 12 months from the start of COS using blastocysts obtained in this trial.

Exclusion Criteria:

* More than one previous COS cycle for IVF/ICSI.
* Known endometriosis stage III-IV (defined by the revised ASRM classification, 2012 ).
* Known history of anovulation.
* One or more follicles greater than or equal to 10 mm (including cysts) observed on the transvaginal ultrasound prior to randomization on stimulation day 1.
* Known history of recurrent miscarriage (defined as three consecutive losses after ultrasound confirmation of pregnancy [excluding ectopic pregnancy] and before week 24 of pregnancy).
* Known abnormal karyotype of participant or of her partner / sperm donor, as applicable, depending on source of sperm used for insemination in this trial. In case partner sperm will be used and the sperm production is severely impaired (concentration <1 million/mL), normal karyotype, including no Y-chromosome microdeletion, must be documented.
* Any known clinically significant systemic disease (e.g. insulin-dependent diabetes).
* Known inherited or acquired thrombophilia.
* Active arterial or venous thromboembolism or severe thrombophlebitis, or a history of these events.
* Any known endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney) with the exception of pharmacologically controlled sub-clinical hypothyroidism.
* Known tumors of the ovary, breast, uterus, adrenal gland, pituitary or hypothalamus which would contraindicate the use of gonadotropins.
* Known moderate or severe impairment of renal or hepatic function.
* Any abnormal finding of clinical chemistry, hematology, thyroid-stimulating hormone (TSH) or prolactin, or vital signs at screening, which is judged clinically significant by the investigator.
* Known abnormal cervical cytology of clinical significance observed within three years prior to randomization (unless the clinical significance has been resolved).
* Findings at the gynecological examination at screening which preclude gonadotropin stimulation or are associated with a reduced chance of pregnancy, e.g. congenital uterine abnormalities or retained intrauterine device.
* Pregnancy (negative urinary pregnancy tests must be documented at screening and prior to randomization) or contraindication to pregnancy.
* Known current active pelvic inflammatory disease.
* Use of fertility modifiers during the last menstrual cycle before randomization, including dehydroepiandrosterone (DHEA), metformin or cycle programming with oral contraceptives, progestogen or estrogen preparations.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pre-menopausal females between the ages of 18 and 34 years at the time of randomization.
Enrollment: 579 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (23):
- United States (23):
  - Fertility Treatment Center, Tempe, Arizona
  - HRC Fertility, Encino, California
  - Center for Advanced Reproductive Services PC, Farmington, Connecticut
  - Reproductive Associates of Delaware, Newark, Delaware
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Center for Reproductive Medicine, Winter Park, Florida
  - Fertility Institute of Hawaii, INC, Honolulu, Hawaii
  - Fertility Centers of Illinois (RH), Chicago, Illinois
  - InVia Fertility, Hoffman Estates, Illinois
  - Boston IVF, Waltham, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Reproductive Endocrinology Associates of Charlotte (REACH) S. Corporation, Charlotte, North Carolina
  - Carolina Conceptions, Raleigh, North Carolina
  - Institute for Reproductive Health, Cincinnati, Ohio
  - Abington Reproductive Medicine, Abington, Pennsylvania
  - Main Line Fertility Center, Bryn Mawr, Pennsylvania
  - Fertility Associates of Memphis, PLLC, Memphis, Tennessee
  - Center for Assisted Reproduction, Bedford, Texas
  - Houston Fertility Institute, Houston, Texas
  - Center of Reproductive Medicine, Webster, Texas
  - Utah Fertility Center, Pleasant Grove, Utah
  - Eastern Virginia Medical School | EVMS Obstetrics & Gynecology, Norfolk, Virginia
  - Seattle Reproductive Medicine WA, Seattle, Washington

REFERENCES:
- [Derived] Scheiber MD, Doody KJ, Foster ED, Grover SA, Heiser PW; RITA-1 and RITA-2 (Recombinant FSH Investigation in the Treatment of Infertility with ART) trial groups. Ovarian stimulation with follitropin delta is safe and effective: results from the RITA randomized, double-blind, placebo-controlled trials. Fertil Steril. 2026 Jan;125(1):54-63. doi: 10.1016/j.fertnstert.2025.07.032. Epub 2025 Jul 24. PMID 40714031

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed in 23 investigational sites in 17 states of the United States between Oct 2018 to Nov 2020.
Pre-assignment Details: In total, 647 participants were screened of which 579 participants were randomized. Of the randomized participants, 578 participants were exposed to the investigational medicinal product (IMP): 525 to FE 999049 (Follitropin Delta) and 53 to Placebo. One participant was randomization failure and did not receive the IMP.
Groups:
- FE 999049 (Follitropin Delta): FE 999049 was administered as single daily subcutaneous injections in the abdomen at a starting dose of 12 µg daily that was fixed for the first four stimulation days. Based on ovarian response, the dose could be adjusted by 3 µg, with dose increases implemented not more frequently than once every 2 days and dose decreases implemented per investigator's judgement. The minimum daily dose was 6 µg, and the maximum daily dose was 24 µg.
  Participants could be treated for a maximum of 20 days. Coasting, use of dopamine agonist or any other drug to prevent early ovarian hyperstimulation syndrome (OHSS) with the exception of gonadotropin-releasing hormone (GnRH) agonist for triggering of final follicular maturation, was not allowed.
Period: Overall Study
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Started (This trial assessed the efficacy and safety of FE 999049 in participants undergoing controlled ovarian stimulation (COS) for in-vitro fertilization (IVF) / intracytoplasmic sperm injection (ICSI) following a GnRH antagonist protocol. The trial was designed to capture the clinical efficacy of a single COS cycle in a more complete manner by following outcomes from both the fresh and subsequent cryopreserved cycles.) | 526 | 53
mITT | 525 | 53
Completed | 506 | 52
Not Completed | 20 | 1
Not completed — Protocol deviation | 13 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Randomization failure | 1 | 0
Not completed — Participant withdrew consent | 1 | 0
Not completed — Participant withdrew from trial | 2 | 1

BASELINE CHARACTERISTICS:
Population: The modified intention-to-treat (mITT) analysis set comprised all randomized and exposed participants. Participants were analyzed according to planned treatment.
Groups:
- FE 999049 (Follitropin Delta): FE 999049 was administered as single daily subcutaneous injections in the abdomen at a starting dose of 12 µg daily that was fixed for the first four stimulation days. Based on ovarian response, the dose could be adjusted by 3 µg, with dose increases implemented not more frequently than once every 2 days and dose decreases implemented per investigator's judgement. The minimum daily dose was 6 µg, and the maximum daily dose was 24 µg.
  Participants could be treated for a maximum of 20 days. Coasting, use of dopamine agonist or any other drug to prevent early OHSS with the exception of GnRH agonist for triggering of final follicular maturation, was not allowed.
- Total: Total of all reporting groups
Arm/Group | FE 999049 (Follitropin Delta) | Placebo | Total
Number analyzed (Participants) | 525 | 53 | 578
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (2.7) | 30.9 (2.9) | 30.7 (2.8)
Age, Customized [Count of Participants; unit: Participants]
  18-24 years | 16 | 2 | 18
  25-29 years | 147 | 16 | 163
  30-34 years | 362 | 35 | 397
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 525 | 53 | 578
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 6 | 66
  Not Hispanic or Latino | 465 | 47 | 512
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 33 | 6 | 39
  Native Hawaiian or Other Pacific Islander | 5 | 0 | 5
  Black or African American | 49 | 2 | 51
  White | 437 | 45 | 482
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (5.1) | 26.5 (4.8) | 26.5 (5.1)
Primary infertility [Count of Participants; unit: Participants] | 318 | 29 | 347
Duration of infertility (months) [Mean (Standard Deviation); unit: months] | 36.5 (25.4) | 38.2 (18.3) | 36.6 (24.8)
Primary reason for infertility [Count of Participants; unit: Participants]
  Unexplained infertility | 234 | 22 | 256
  Tubal infertility | 83 | 6 | 89
  Mild male factor | 54 | 3 | 57
  Moderate male factor | 81 | 6 | 87
  Severe male factor | 49 | 11 | 60
  Endometriosis stage I/II | 24 | 5 | 29

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Ongoing Pregnancy Rate After the Fresh Cycle and Cryopreserved Cycles Initiated Within 12 Months From the Start of COS
Description: Defined as at least one intrauterine viable fetus 8-9 weeks after transfer. Data in this endpoint are presented for the fresh cycle and the cryopreserved cycles.
Time Frame: 8-9 weeks after transfer (up to approximately 16 months after start of stimulation)
Population: The mITT analysis set comprised all randomized and exposed participants. Participants were analyzed according to planned treatment.
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants | 63.0 | 0.0
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs Placebo; Test type: Other; p < 0.001, Fisher Exact; Treatment difference = 63.0, 95% CI 2-sided [55.5 to 67.1] — 95% exact Agresti-Min confidence intervals

2. Secondary Outcome: Ongoing Pregnancy Rate in the Fresh Cycle and in the Cryopreserved Cycles
Description: as for outcome 1
Time Frame: 8-9 weeks after transfer (up to approximately 16 months after start of stimulation)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants
  Fresh cycle | 29.5 | 0.0
  Cryopreserved cycles: number analyzed (Participants) | 278 | 53
  Cryopreserved cycles | 65.8 | 0
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs Placebo; Ongoing Pregnancy Rate in the Fresh Cycle; Test type: Other; p < 0.001, Fisher Exact; Treatment difference = 29.5, 95% CI 2-sided [22.5 to 33.7] — 95% exact Agresti-Min confidence intervals

3. Secondary Outcome: Time From Start of COS to Ongoing Pregnancy Across the Fresh and Cryopreserved Cycles
Description: Time from start of COS to ongoing pregnancy, including both the fresh and cryopreserved cycles.
  In the placebo group, no participants achieved an ongoing pregnancy either after 12 calendar months or after 12 study months.
Time Frame: 8-9 weeks after transfer (up to approximately 16 months after start of stimulation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 525
days
  Total number of days until ongoing pregnancy 12 study months | 133.0 (82.5)
  Total number of days until ongoing pregnancy 12 calendar months | 127.6 (70.0)

4. Secondary Outcome: Time From Start of COS to Ongoing Pregnancy Across the Fresh and Cryopreserved Cycles, Measured in Number of Cycles Before Achieving Ongoing Pregnancy
Description: Time from start of COS to ongoing pregnancy, including both the fresh and cryopreserved cycles, measured in number of cycles before achieving ongoing pregnancy.
  In the placebo group, no participants achieved an ongoing pregnancy either after 12 calendar months or after 12 study months.
Time Frame: 8-9 weeks after transfer (up to approximately 16 months after start of stimulation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cycles
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 336
Cycles
  Number of cycles until ongoing pregnancy 12 study months | 1.8 (0.9)
  Number of cycles until ongoing pregnancy 12 calendar months: number analyzed (Participants) | 331
  Number of cycles until ongoing pregnancy 12 calendar months | 1.8 (0.9)

5. Secondary Outcome: Ongoing Implantation Rate in the Fresh Cycle, the Cryopreserved Cycles and Cumulatively
Description: Defined as the number of intrauterine viable fetuses 8-9 weeks after transfer divided by number of blastocysts transferred. Data in this endpoint are presented for the fresh cycle, the cryopreserved cycles, and all cycles.
  One participant can contribute with a range from zero to multiple blastocysts.
  Data is not shown for placebo arm because no blastocyst transfer was performed in the fresh cycle or cryopreserved cycles.
  '%' in the unit of measure refers to 'percentage'.
Time Frame: 8-9 weeks after transfer (up to approximately 16 months after start of stimulation)
Population: as for outcome 1
Measure: Number; unit: % of viable fetus/blastocyst transfer
Units Other Than Participants: Blastocysts
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 525
Number analyzed (Blastocysts) | 729
% of viable fetus/blastocyst transfer
  Fresh cycle: number analyzed (Blastocysts) | 313
  Fresh cycle | 49.5
  Cryopreserved cycles: number analyzed (Blastocysts) | 416
  Cryopreserved cycles | 44.2
  All cycles | 46.5

6. Secondary Outcome: Clinical Pregnancy Rate in the Fresh Cycle, the Cryopreserved Cycles and Cumulatively
Description: Defined at least one gestational sac 5-6 weeks after transfer. Data in this endpoint are presented for the fresh cycle, the cryopreserved cycles, and all cycles.
Time Frame: 5-6 weeks after transfer (up to approximately 15 months after start of stimulation)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants
  Fresh cycle | 31.8 | 0
  Cryopreserved cycles: number analyzed (Participants) | 278 | 53
  Cryopreserved cycles | 72.3 | 0
  All cycles | 68.2 | 0
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs Placebo; Clinical pregnancy rate in the fresh cycle; Test type: Other; p < 0.001, Fisher Exact; Treatment difference = 31.8, 95% CI 2-sided [24.7 to 36.0] — 95% exact Agresti-Min confidence intervals
Statistical Analysis 2: Comparison: FE 999049 (Follitropin Delta) vs Placebo; Clinical pregnancy rate cumulatively; Test type: Other; p < 0.001, Fisher Exact; Treatment difference = 68.2, 95% CI 2-sided [61.2 to 72.1] — 95% exact Agresti-Min confidence intervals

7. Secondary Outcome: Vital Pregnancy Rate in the Fresh Cycle, the Cryopreserved Cycles and Cumulatively
Description: Defined at least one intrauterine gestational sac with fetal heart beat 5-6 weeks after transfer. Data in this endpoint are presented for the fresh cycle, the cryopreserved cycles, and all cycles.
Time Frame: 5-6 weeks after transfer (up to approximately 15 months after start of stimulation)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants
  Fresh cycle | 30.5 | 0
  Cryopreserved cycles: number analyzed (Participants) | 278 | 53
  Cryopreserved cycles | 67.3 | 0
  All cycles | 65.1 | 0
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs Placebo; Vital pregnancy rate in the fresh cycle; Test type: Other; p < 0.001, Fisher Exact; Treatment difference = 30.5, 95% CI 2-sided [23.4 to 34.6] — 95% exact Agresti-Min confidence intervals
Statistical Analysis 2: Comparison: FE 999049 (Follitropin Delta) vs Placebo; Vital pregnancy rate cumulatively; Test type: Other; p < 0.001, Fisher Exact; Treatment difference = 65.1, 95% CI 2-sided [57.5 to 69.1] — 95% exact Agresti-Min confidence intervals

8. Secondary Outcome: Implantation Rate in the Fresh Cycle, the Cryopreserved Cycles and Cumulatively
Description: Defined as the number of gestational sacs 5-6 weeks after transfer divided by number of blastocysts transferred. Data in this endpoint are presented for the fresh cycle, the cryopreserved cycles, and all cycles.
  One participant can contribute with a range from zero to multiple blastocysts.
  Data is not shown for placebo arm because no subjects underwent blastocyst transfer in the fresh cycle or cryopreserved cycles.
  '%' in the unit of measure refers to 'percentage'.
Time Frame: 5-6 weeks after transfer (up to approximately 15 months after start of stimulation)
Population: as for outcome 1
Measure: Number; unit: % gestational sacs/blastocyst transfer
Units Other Than Participants: Blastocysts
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 525
Number analyzed (Blastocysts) | 729
% gestational sacs/blastocyst transfer
  Fresh cycle: number analyzed (Blastocysts) | 313
  Fresh cycle | 53.4
  Cryopreserved cycles: number analyzed (Blastocysts) | 416
  Cryopreserved cycles | 51.7
  All cycles | 52.4

9. Secondary Outcome: Positive Beta Human Chorionic Gonadotropin (βhCG) Rate in the Fresh Cycle, the Cryopreserved Cycles and Cumulatively
Description: Defined as positive serum βhCG test 10-14 days after transfer. Data in this endpoint are presented for the fresh cycle, the cryopreserved cycles, and all cycles.
Time Frame: 10-14 days after transfer (up to approximately 14 months after start of stimulation)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants
  Fresh cycle | 35.0 | 0
  Cryopreserved cycles: number analyzed (Participants) | 278 | 53
  Cryopreserved cycles | 78.1 | 0
  All cycles | 72.4 | 0
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs Placebo; Positive βhCG rate in the fresh cycle; Test type: Other; p < 0.001, Fisher Exact; Treatment difference = 35.0, 95% CI 2-sided [28.1 to 39.2] — 95% exact Agresti-Min confidence intervals
Statistical Analysis 2: Comparison: FE 999049 (Follitropin Delta) vs Placebo; Positive βhCG rate cumulatively; Test type: Other; p < 0.001, Fisher Exact; Treatment difference = 72.4, 95% CI 2-sided [65.3 to 76.2] — 95% exact Agresti-Min confidence intervals

10. Secondary Outcome: Proportion of Subjects in the Fresh Cycle With Triggering of Final Follicular Maturation (hCG, With GnRH Agonist, and in Total), Cycle Cancellation and Transfer Cancellation
Description: Data in this endpoint are presented for the fresh cycle.
Time Frame: Up to 5 days after oocyte retrieval (up to 27 days after start of stimulation)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- FE 999049 (Follitropin Delta): FE 999049 was administered as single daily subcutaneous injections in the abdomen at a starting dose of 12 µg daily that was fixed for the first four stimulation days. Based on ovarian response, the dose could be adjusted by 3 µg, with dose increases implemented not more frequently than once every 2 days and dose decreases implemented per investigator's judgement. The minimum daily dose was 6 µg, and the maximum daily dose was 24 µg. Transfer cancellation is mandatory in participants undergoing triggering with GnRH agonist and participants with >=20 oocytes retrieved.
  Participants could be treated for a maximum of 20 days. Coasting, use of dopamine agonist or any other drug to prevent early OHSS with the exception of GnRH agonist for triggering of final follicular maturation, was not allowed.
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants
  Triggering drug (hCG) | 77.0 | 1.9
  Triggering drug (GnRH agonist) | 21.5 | 0.0
  Triggering drug (None) | 1.5 | 98.1
  Cycle cancellation | 1.5 | 98.1
  Transfer cancellation | 38.9 | 1.9

11. Secondary Outcome: Number of Follicles on Stimulation Day 5
Description: The total number of follicles and the number of follicles per size category are presented
Time Frame: On stimulation day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of follicles
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
number of follicles
  Total number of follicles | 19.3 (9.9) | 16.5 (7.1)
  Follicles >= 12 mm | 1.7 (2.0) | 0.3 (0.7)
  Follicles >= 17 mm | 0.0 (0.2) | 0.0 (0.0)

12. Secondary Outcome: Number of Follicles at End-of-stimulation
Description: The total number of follicles and the number of follicles per size category is reported.
Time Frame: At end-of-stimulation (up to 20 stimulation days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of follicles
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 524 | 53
number of follicles
  Total number of follicles | 23.0 (11.8) | 15.6 (7.6)
  Follicles >= 12 mm | 13.0 (7.3) | 0.7 (0.5)
  Follicles >= 17 mm | 4.4 (2.5) | 0.3 (0.5)

13. Secondary Outcome: Size of Follicles on Stimulation Day 5
Description: Counted by ultrasound for the right and left ovary for each participant.
Time Frame: On stimulation day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
mm
  Largest follicle (mm) | 12.2 (2.0) | 9.9 (2.4)
  Average size of 2 largest follicles (mm) | 11.7 (1.8) | 9.2 (2.0)

14. Secondary Outcome: Size of Follicles at End-of-stimulation
Description: Counted by ultrasound for the right and left ovary for each participant.
Time Frame: At end-of-stimulation (up to 20 stimulation days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 524 | 53
mm
  Largest follicle (mm) | 19.9 (2.0) | 13.6 (4.8)
  Average size of 2 largest follicles (mm) | 19.2 (1.6) | 10.9 (2.8)

15. Secondary Outcome: Number of Oocytes Retrieved
Description: The number of oocytes retrieved was recorded at the oocyte retrieval visit.
Time Frame: On day of oocyte retrieval (up to 22 days after start of stimulation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of oocytes retrieved
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
number of oocytes retrieved | 15.1 (10.4) | 0.0 (0.0)

16. Secondary Outcome: Proportion of Subjects With <4, 4-7, 8-14, 15-19 and ≥20 Oocytes Retrieved
Description: Grouped according to the number of oocytes retrieved. Participants with cycle cancellation due to poor ovarian response are included in the <4 oocytes group.
Time Frame: On day of oocyte retrieval (up to 22 days after start of stimulation)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants
  <4 oocytes retrieved | 6.7 | 100
  4-7 oocytes retrieved | 13.9 | 0
  8-14 oocytes retrieved | 36.6 | 0
  15-19 oocytes retrieved | 18.7 | 0
  >=20 oocytes retrieved | 24.2 | 0

17. Secondary Outcome: Number of Metaphase II Oocytes
Description: The number of MII oocytes to oocytes retrieved for participants where all oocytes were inseminated using ICSI are presented.
Time Frame: On day of oocyte retrieval (up to 22 days after start of stimulation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of MII oocytes
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 427
number of MII oocytes | 10.9 (7.6)

18. Secondary Outcome: Number of Fertilized Oocytes
Description: An oocyte was defined as fertilized if it had 2 pronuclei (2PN) at 19h (±2h).
Time Frame: On day 1 after oocyte retrieval (up to 23 days after start of stimulation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: oocytes (number of fertilized oocytes)
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
oocytes (number of fertilized oocytes) | 8.4 (6.3) | 0.0 (0.0)

19. Secondary Outcome: Fertilization Rate
Description: The fertilization rate was defined as the number of 2PN oocytes divided by the number of oocytes retrieved.
  Fertilization rate relative to oocytes retrieved has been reported.
  Data is not shown for placebo arm because the mean number of fertilized oocytes was 0 in all subjects, since no subjects had oocytes retrieved or fertilized.
Time Frame: On day 1 after oocyte retrieval (up to 23 days after start of stimulation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of fertilized oocytes
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 515
percentage of fertilized oocytes | 56.6 (21.3)

20. Secondary Outcome: Number and Quality of Blastocysts on Day 5 After Oocyte Retrieval
Description: Number of blastocysts (total and good-quality) on Day 5 are presented. The quality evaluation of blastocysts consisted of assessment of three parameters, as per the Gardner & Schoolcraft system: blastocyst expansion and hatching status (graded: 1-6), inner cell mass (graded: A-D) and trophectoderm (graded: A-D). A good-quality blastocyst was defined as a blastocyst of grade 3BB or higher.
Time Frame: On day 5 after oocyte retrieval
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: blastocysts
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
blastocysts
  Number of blastocysts on day 5 | 5.0 (4.3) | 0.0 (0.0)
  Number of good-quality blastocysts on day 5 | 3.4 (3.3) | 0.0 (0.0)

21. Secondary Outcome: Endometrial Thickness on Stimulation Day 5
Description: Mean endometrial thickness is reported.
Time Frame: On stimulation day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
mm | 8.2 (2.1) | 5.8 (1.8)
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs Placebo; Test type: Other; p < 0.001, Wilcoxon rank sum test

22. Secondary Outcome: Endometrial Thickness at End-of-stimulation
Description: Mean endometrial thickness is reported.
Time Frame: At end-of-stimulation (up to 20 stimulation days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 524 | 53
mm | 10.9 (2.3) | 7.5 (2.2)
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs Placebo; Test type: Other; p < 0.001, Wilcoxon rank sum test

23. Secondary Outcome: Echogenicity Pattern on Stimulation Day 5
Description: The distribution of participants with hypoechogenic, isoechogenic, or hyperechogenic endometrium is reported.
Time Frame: On stimulation day 5
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants
  Hypoechogenic | 66.7 | 58.5
  Isoechogenic | 2.9 | 7.5
  Hyperechogenic | 29.9 | 34.0
  Not possible to evaluate | 0.6 | 0
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs Placebo; Test type: Other; p = 0.220, Fisher Exact

24. Secondary Outcome: Echogenicity Pattern at End-of-stimulation
Description: The distribution of participants with hypoechogenic, isoechogenic, or hyperechogenic endometrium is reported.
Time Frame: At end-of-stimulation (up to 20 stimulation days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 524 | 53
percentage of participants
  Hypoechogenic | 68.1 | 64.2
  Isoechogenic | 3.1 | 5.7
  Hyperechogenic | 28.4 | 30.2
  Not possible to evaluate | 0.4 | 0
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs Placebo; Test type: Other; p = 0.588, Fisher Exact

25. Secondary Outcome: Oocyte Utilization Rate
Description: Defined as the number of blastocysts transferred or cryopreserved divided by the number of oocytes retrieved.
  Data in this endpoint are presented for the cryopreserved cycles.
Time Frame: On day of oocyte retrieval up to 12 months after start of COS
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: blastocysts/oocyte retrieved
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 515
blastocysts/oocyte retrieved | 31.6 (20.6)

26. Secondary Outcome: Oocyte Efficiency Index
Description: Defined as the cumulative number of ongoing pregnancies per oocyte retrieved.
  Data in this endpoint are presented for the cryopreserved cycles.
  The unit of measure for this endpoint is 'cumulative ongoing pregnancies/oocyte retrieved'.
Time Frame: 8-9 weeks after transfer
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ongoing pregnancies/oocyte retrieved
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 515
ongoing pregnancies/oocyte retrieved | 5.8 (6.9)

27. Secondary Outcome: Percentage of Blastocysts Surviving Cryopreservation
Description: Data in this endpoint are presented for the cryopreserved cycles.
  The unit is number of blastocysts with observations. One participant can contribute with a range from zero to multiple blastocysts.
Time Frame: 0 hour (+0.5 hour) after thawing
Population: as for outcome 1
Measure: Number; unit: percentage of blastocysts
Units Other Than Participants: Number of blastocyst warmed
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 525
Number analyzed (Number of blastocyst warmed) | 421
percentage of blastocysts | 98.8

28. Secondary Outcome: Percentage of Blastocysts With Re-expansion After Cryopreservation
Description: as for outcome 27
Time Frame: 2.5 hour (±0.5 hour) after thawing
Population: as for outcome 1
Measure: Number; unit: percentage of blastocysts
Units Other Than Participants: Number of blastocyst warmed
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 525
Number analyzed (Number of blastocyst warmed) | 421
percentage of blastocysts | 97.1

29. Secondary Outcome: Number of Cryopreserved Cycles Initiated Within 12 Months From the Start of COS
Description: The total number of cryopreserved cycles initiated are reported.
  One participant can contribute with multiple cycles.
  Data in this endpoint are presented for the cryopreserved cycles.
Time Frame: Up to 12 months after start of stimulation
Population: as for outcome 1
Measure: Number; unit: cycles
Units Other Than Participants: Cryopreserved cycles initiated
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 278
Number analyzed (Cryopreserved cycles initiated) | 466
cycles
  Programmed cycles initiated | 423
  Natural cycles initiated | 43

30. Secondary Outcome: Number of Cryopreserved Cycles With Blastocyst Transfer
Description: The total number of cryopreserved cycles with blastocyst transfer are reported.
  One participant can contribute with multiple cycles.
  Data in this endpoint are presented for the cryopreserved cycles.
Time Frame: Up to 12 months after start of stimulation
Population: as for outcome 1
Measure: Number; unit: cycles
Units Other Than Participants: Cryopreserved cycles with transfer
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 278
Number analyzed (Cryopreserved cycles with transfer) | 416
cycles
  Programmed cycles with transfer | 380
  Natural cycles with transfer | 36

31. Secondary Outcome: Circulating Concentrations of Anti-mullerian Hormone (AMH)
Description: Blood samples for analysis of circulating concentrations of AMH were drawn. The median and inter-quartile range (IQR) of AMH levels on stimulation day 1, stimulation day 5, end-of-stimulation visit and oocyte retrieval visit are presented.
Time Frame: From screening to the day of oocyte retrieval (up to 22 days after start of stimulation)
Population: The mITT analysis set comprised all randomized and exposed participants. Participants were analyzed according to planned treatment.
  No circulating concentrations of AMH were assessed for the oocyte retrieval visit for the placebo arm, because no participants who received placebo became pregnant.
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 524 | 53
pmol/L
  Stimulation day 1 | 20.7 [12.9 to 31.3] | 18.5 [13.9 to 26.7]
  Stimulation day 5: number analyzed (Participants) | 515 | 51
  Stimulation day 5 | 17.6 [10.7 to 26.3] | 20.4 [13.3 to 27.5]
  End-of-stimulation visit: number analyzed (Participants) | 506 | 48
  End-of-stimulation visit | 10.4 [6.6 to 15.9] | 20.9 [14.6 to 31.3]
  Oocyte retrieval visit: number analyzed (Participants) | 505 | 0
  Oocyte retrieval visit | 7.9 [5.2 to 12.2] |

32. Secondary Outcome: Circulating Concentrations of Follicle-stimulating Hormone (FSH)
Description: Blood samples for analysis of circulating concentrations of FSH were drawn. The median and IQR of FSH levels on stimulation day 1, stimulation day 5, end-of-stimulation visit and oocyte retrieval visit are presented.
Time Frame: From screening to the day of oocyte retrieval (up to 22 days after start of stimulation)
Population: The mITT analysis set comprised all randomized and exposed participants. Participants were analyzed according to planned treatment.
  No circulating concentrations of FSH were assessed for the oocyte retrieval visit for the placebo arm, because no participants who received placebo became pregnant.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 520 | 53
IU/L
  Stimulation day 1 | 8.3 [7.1 to 9.7] | 8.5 [7.6 to 10.3]
  Stimulation day 5 | 16.9 [14.2 to 20.1] | 8.2 [7.3 to 9.2]
  End-of-stimulation visit: number analyzed (Participants) | 517 | 47
  End-of-stimulation visit | 20.8 [16.5 to 25.1] | 6.7 [5.2 to 8.4]
  Oocyte retrieval visit: number analyzed (Participants) | 505 | 0
  Oocyte retrieval visit | 11.7 [9.9 to 14.5] |

33. Secondary Outcome: Circulating Concentrations of Luteinizing Hormone (LH)
Description: Blood samples for analysis of circulating concentrations of LH were drawn. The median and IQR of LH levels on stimulation day 1, stimulation day 5, end-of-stimulation visit and oocyte retrieval visit are presented.
Time Frame: From screening to the day of oocyte retrieval (up to 22 days after start of stimulation)
Population: The mITT analysis set comprised all randomized and exposed participants. Participants were analyzed according to planned treatment.
  No circulating concentrations of LH were assessed for the oocyte retrieval visit for the placebo arm, because no participants who received placebo became pregnant.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 522 | 53
IU/L
  Stimulation day 1 | 5.1 [3.8 to 6.6] | 4.7 [3.9 to 5.5]
  Stimulation day 5: number analyzed (Participants) | 520 | 53
  Stimulation day 5 | 2.2 [1.6 to 3.2] | 6.0 [4.9 to 7.4]
  End-of-stimulation visit: number analyzed (Participants) | 518 | 48
  End-of-stimulation visit | 1.9 [1.1 to 3.1] | 7.7 [6.0 to 10.6]
  Oocyte retrieval visit: number analyzed (Participants) | 502 | 0
  Oocyte retrieval visit | 2.2 [1.1 to 3.7] |

34. Secondary Outcome: Circulating Concentrations of Estradiol
Description: Blood samples for analysis of circulating concentrations of estradiol were drawn. The median and IQR of estradiol levels on stimulation day 1, stimulation day 5, end-of-stimulation visit and oocyte retrieval visit are presented.
Time Frame: From screening to the day of oocyte retrieval (up to 22 days after start of stimulation)
Population: The mITT analysis set comprised all randomized and exposed participants. Participants were analyzed according to planned treatment.
  No circulating concentrations of estradiol were assessed for the oocyte retrieval visit for the placebo arm, because no participants who received placebo became pregnant.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 522 | 53
pg/mL
  Stimulation day 1 | 39.5 [32.8 to 48.7] | 37.7 [31.7 to 50.8]
  Stimulation day 5: number analyzed (Participants) | 520 | 53
  Stimulation day 5 | 404.1 [255.4 to 624.2] | 53.6 [42.1 to 75.6]
  End-of-stimulation visit: number analyzed (Participants) | 515 | 48
  End-of-stimulation visit | 1846.9 [1122.1 to 2729.5] | 105.5 [58.3 to 163.6]
  Oocyte retrieval visit: number analyzed (Participants) | 511 | 0
  Oocyte retrieval visit | 931.2 [570.0 to 1475.8] |

35. Secondary Outcome: Circulating Concentrations of Progesterone
Description: Blood samples for analysis of circulating concentrations of progesterone were drawn. The median and IQR of progesterone levels on stimulation day 1, stimulation day 5, end-of-stimulation visit and oocyte retrieval visit are presented.
Time Frame: From screening to the day of oocyte retrieval (up to 22 days after start of stimulation)
Population: The mITT analysis set comprised all randomized and exposed participants. Participants were analyzed according to planned treatment.
  No circulating concentrations of progesterone were assessed for the oocyte retrieval visit for the placebo arm, because no participants who received placebo became pregnant.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 522 | 53
ng/mL
  Stimulation day 1 | 0.6 [0.3 to 0.8] | 0.5 [0.3 to 0.7]
  Stimulation day 5: number analyzed (Participants) | 520 | 53
  Stimulation day 5 | 0.6 [0.3 to 0.8] | 0.5 [0.3 to 0.7]
  End-of-stimulation visit: number analyzed (Participants) | 518 | 48
  End-of-stimulation visit | 1.1 [0.8 to 1.5] | 0.5 [0.3 to 0.6]
  Oocyte retrieval visit: number analyzed (Participants) | 502 | 0
  Oocyte retrieval visit | 6.7 [4.6 to 9.9] |

36. Secondary Outcome: Circulating Concentrations of Inhibin A
Description: Blood samples for analysis of circulating concentrations of inhibin A were drawn. The median and IQR of inhibin A levels on stimulation day 1, stimulation day 5, end-of-stimulation visit and oocyte retrieval visit are presented.
Time Frame: From screening to the day of oocyte retrieval (up to 22 days after start of stimulation)
Population: The mITT analysis set comprised all randomized and exposed participants. Participants were analyzed according to planned treatment.
  No circulating concentrations of Inhibin A were assessed for the oocyte retrieval visit for the placebo arm, because no participants who received placebo became pregnant.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 514 | 52
pg/mL
  Stimulation day 1 | 4.3 [2.8 to 6.0] | 4.3 [3.4 to 5.0]
  Stimulation day 5: number analyzed (Participants) | 512 | 51
  Stimulation day 5 | 71.3 [46.9 to 110.8] | 7.3 [4.5 to 10.0]
  End-of-stimulation visit: number analyzed (Participants) | 507 | 48
  End-of-stimulation visit | 329.8 [226.9 to 480.4] | 12.4 [7.7 to 22.6]
  Oocyte retrieval visit: number analyzed (Participants) | 502 | 0
  Oocyte retrieval visit | 255.6 [180.5 to 370.2] |

37. Secondary Outcome: Circulating Concentrations of Inhibin B
Description: Blood samples for analysis of circulating concentrations of inhibin B were drawn. The median and IQR of inhibin B levels on stimulation day 1, stimulation day 5, end-of-stimulation visit and oocyte retrieval visit are presented.
Time Frame: From screening to the day of oocyte retrieval (up to 22 days after start of stimulation)
Population: The mITT analysis set comprised all randomized and exposed participants. Participants were analyzed according to planned treatment.
  No circulating concentrations of Inhibin B were assessed for the oocyte retrieval visit for the placebo arm, because no participants who received placebo became pregnant.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 516 | 52
pg/mL
  Stimulation day 1 | 82.0 [61.0 to 104.0] | 80.0 [58.5 to 104.5]
  Stimulation day 5: number analyzed (Participants) | 509 | 51
  Stimulation day 5 | 682.0 [453.0 to 955.0] | 105.0 [82.0 to 129.0]
  End-of-stimulation visit: number analyzed (Participants) | 504 | 48
  End-of-stimulation visit | 1106.0 [665.0 to 1640.0] | 79.5 [59.0 to 111.5]
  Oocyte retrieval visit: number analyzed (Participants) | 499 | 0
  Oocyte retrieval visit | 445.0 [266.0 to 675.0] |

38. Secondary Outcome: Total Gonadotropin Dose
Description: Calculated by start dates, end dates and daily dose of IMP.
Time Frame: Up to 20 stimulation days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram of dose
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
microgram of dose | 104.2 (25.3) | 115.9 (19.1)

39. Secondary Outcome: Number of Stimulation Days
Description: Calculated by start dates and end dates.
Time Frame: Up to 20 stimulation days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
days | 8.1 (1.4) | 8.3 (0.8)

40. Secondary Outcome: Proportion of Participants With Investigator-requested Gonadotropin Dose Adjustments
Description: Investigator-requested decreases and increases of the gonadotropin dose.
Time Frame: Stimulation Day 5
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants
  Decrease | 6.3 | 0
  No change | 55.8 | 20.8
  Increase | 37.9 | 79.2

41. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: Any AE occurring after start of IMP and before the end-of-trial visit, or a pre-treatment AE or pre-existing medical condition that worsens in intensity after start of IMP and before the end-of-trial visit was considered treatment-emergent, and is presented for this endpoint.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From time of signing informed consent until the end-of-cycle visit in the fresh cycle (up to approximately 6 months)
Population: The safety analysis set comprised all randomized and exposed participants. Participants were analyzed according to actual treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants | 54.7 | 9.4

42. Secondary Outcome: Intensity of AEs
Description: The intensity of AE was classified using the following 3-point scale: mild = awareness of signs or symptoms, but no disruption of usual activity; moderate = event sufficient to affect usual activity (disturbing); or severe = inability to work or perform usual activities (unacceptable).
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From time of signing informed consent until the end-of-cycle visit in the fresh cycle (up to approximately 6 months)
Population: as for outcome 41
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants
  Mild AEs | 47.0 | 9.4
  Moderate AEs | 16.6 | 0.0
  Severe AEs | 1.0 | 0.0

43. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Compared to Baseline: Albumin, Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameters including: Albumin and protein.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 513 | 51
g/L
  Albumin (End-of-stimulation visit): number analyzed (Participants) | 513 | 47
  Albumin (End-of-stimulation visit) | -1.68 (2.37) | 0.21 (3.04)
  Albumin (End-of-cycle visit): number analyzed (Participants) | 504 | 51
  Albumin (End-of-cycle visit) | -2.03 (2.92) | -0.29 (2.63)
  Protein (End-of-stimulation visit): number analyzed (Participants) | 512 | 47
  Protein (End-of-stimulation visit) | -3.07 (3.83) | -0.02 (4.35)
  Protein (End-of-cycle visit): number analyzed (Participants) | 501 | 51
  Protein (End-of-cycle visit) | -2.06 (4.20) | -0.16 (3.87)

44. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Compared to Baseline: Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase and Gamma Glutamyl Transferase
Description: Blood samples were collected for the analysis of clinical chemistry parameters including: Alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase and gamma glutamyl transferase.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 512 | 51
IU/L
  Alanine aminotransferase (End-of-stimulation visit): number analyzed (Participants) | 495 | 43
  Alanine aminotransferase (End-of-stimulation visit) | -0.5 (7.7) | 2.2 (8.5)
  Alanine aminotransferase (End-of-cycle visit): number analyzed (Participants) | 494 | 50
  Alanine aminotransferase (End-of-cycle visit) | -1.2 (8.6) | 0.5 (4.4)
  Alkaline phosphatase (End-of-stimulation visit): number analyzed (Participants) | 512 | 47
  Alkaline phosphatase (End-of-stimulation visit) | -1.9 (7.1) | 0.6 (6.6)
  Alkaline phosphatase (End-of-cycle visit): number analyzed (Participants) | 501 | 51
  Alkaline phosphatase (End-of-cycle visit) | 0.0 (10.2) | -0.3 (6.1)
  Aspartate aminotransferase (End-of-stimulation visit): number analyzed (Participants) | 493 | 43
  Aspartate aminotransferase (End-of-stimulation visit) | -0.9 (5.9) | 0.6 (3.8)
  Aspartate aminotransferase (End-of-cycle visit): number analyzed (Participants) | 493 | 50
  Aspartate aminotransferase (End-of-cycle visit) | -0.9 (7.1) | -0.1 (3.8)
  Gamma glutamyl transferase (End-of-stimulation visit): number analyzed (Participants) | 512 | 47
  Gamma glutamyl transferase (End-of-stimulation visit) | -1.0 (6.6) | -0.4 (6.5)
  Gamma glutamyl transferase (End-of-cycle visit): number analyzed (Participants) | 501 | 51
  Gamma glutamyl transferase (End-of-cycle visit) | 0.2 (7.8) | 1.4 (6.2)

45. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Compared to Baseline: Bicarbonate, Blood Urea Nitrogen, Calcium, Chloride, Cholesterol, Glucose, Phosphate, Potassium and Sodium
Description: Blood samples were collected for the analysis of clinical chemistry parameters including: Bicarbonate, blood urea nitrogen, calcium, chloride, cholesterol, glucose, phosphate, potassium and sodium.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 514 | 52
mmol/L
  Bicarbonate (End-of-stimulation visit): number analyzed (Participants) | 491 | 43
  Bicarbonate (End-of-stimulation visit) | 0.13 (2.04) | -0.20 (1.85)
  Bicarbonate (End-of-cycle visit): number analyzed (Participants) | 493 | 49
  Bicarbonate (End-of-cycle visit) | -0.88 (2.63) | -0.65 (2.02)
  Blood urea nitrogen (End-of-stimulation visit): number analyzed (Participants) | 512 | 47
  Blood urea nitrogen (End-of-stimulation visit) | -0.3 (1.0) | 0.3 (1.1)
  Blood urea nitrogen (End-of-cycle visit): number analyzed (Participants) | 501 | 51
  Blood urea nitrogen (End-of-cycle visit) | -0.3 (1.2) | 0.1 (1.0)
  Calcium (End-of-stimulation visit): number analyzed (Participants) | 512 | 47
  Calcium (End-of-stimulation visit) | -0.02 (0.09) | 0.01 (0.08)
  Calcium (End-of-cycle visit): number analyzed (Participants) | 501 | 51
  Calcium (End-of-cycle visit) | -0.01 (0.10) | 0.01 (0.10)
  Chloride (End-of-stimulation visit): number analyzed (Participants) | 512 | 47
  Chloride (End-of-stimulation visit) | -0.5 (2.3) | -0.1 (2.1)
  Chloride (End-of-cycle visit): number analyzed (Participants) | 501 | 51
  Chloride (End-of-cycle visit) | 0.4 (2.4) | 0.4 (2.3)
  Cholesterol (End-of-stimulation visit): number analyzed (Participants) | 514 | 47
  Cholesterol (End-of-stimulation visit) | -0.3 (0.5) | 0.1 (0.5)
  Cholesterol (End-of-cycle visit): number analyzed (Participants) | 504 | 52
  Cholesterol (End-of-cycle visit) | 0.2 (0.6) | 0.0 (0.5)
  Glucose (End-of-stimulation visit): number analyzed (Participants) | 495 | 43
  Glucose (End-of-stimulation visit) | -0.2 (0.8) | -0.1 (1.1)
  Glucose (End-of-cycle visit): number analyzed (Participants) | 493 | 50
  Glucose (End-of-cycle visit) | 0.0 (0.9) | -0.2 (0.8)
  Phosphate (End-of-stimulation visit): number analyzed (Participants) | 513 | 47
  Phosphate (End-of-stimulation visit) | -0.05 (0.17) | -0.02 (0.14)
  Phosphate (End-of-cycle visit): number analyzed (Participants) | 504 | 51
  Phosphate (End-of-cycle visit) | 0.02 (0.18) | -0.01 (0.18)
  Potassium (End-of-stimulation visit): number analyzed (Participants) | 512 | 47
  Potassium (End-of-stimulation visit) | 0.00 (0.41) | 0.01 (0.45)
  Potassium (End-of-cycle visit): number analyzed (Participants) | 501 | 51
  Potassium (End-of-cycle visit) | 0.10 (0.49) | 0.13 (0.46)
  Sodium (End-of-stimulation visit): number analyzed (Participants) | 512 | 47
  Sodium (End-of-stimulation visit) | -0.5 (2.2) | 0.4 (2.2)
  Sodium (End-of-cycle visit): number analyzed (Participants) | 501 | 51
  Sodium (End-of-cycle visit) | -0.3 (2.8) | 0.0 (2.4)

46. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Compared to Baseline: Direct Bilirubin, Total Bilirubin, Creatinine, Urate
Description: Blood samples were collected for the analysis of clinical chemistry parameters including: Direct bilirubin, total bilirubin, creatinine, urate.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 512 | 51
umol/L
  Direct bilirubin (End-of-stimulation visit): number analyzed (Participants) | 440 | 39
  Direct bilirubin (End-of-stimulation visit) | -0.01 (0.85) | -0.02 (0.77)
  Direct bilirubin (End-of-cycle visit): number analyzed (Participants) | 475 | 50
  Direct bilirubin (End-of-cycle visit) | -0.26 (0.89) | 0.03 (0.60)
  Total bilirubin (End-of-stimulation visit): number analyzed (Participants) | 493 | 43
  Total bilirubin (End-of-stimulation visit) | -0.26 (2.99) | -0.68 (2.62)
  Total bilirubin (End-of-cycle visit): number analyzed (Participants) | 494 | 50
  Total bilirubin (End-of-cycle visit) | -1.19 (3.85) | 0.03 (2.62)
  Creatinine (End-of-stimulation visit): number analyzed (Participants) | 512 | 47
  Creatinine (End-of-stimulation visit) | -3.50 (7.43) | 1.32 (6.11)
  Creatinine (End-of-cycle visit): number analyzed (Participants) | 501 | 51
  Creatinine (End-of-cycle visit) | -3.11 (10.22) | 2.60 (8.53)
  Urate (End-of-stimulation visit): number analyzed (Participants) | 512 | 47
  Urate (End-of-stimulation visit) | -7.48 (39.36) | -1.52 (30.92)
  Urate (End-of-cycle visit): number analyzed (Participants) | 501 | 51
  Urate (End-of-cycle visit) | -15.04 (51.28) | 14.70 (43.71)

47. Secondary Outcome: Changes in Circulating Levels of Clinical Chemistry Compared to Baseline: Lactate Dehydrogenase
Description: Blood samples were collected for the analysis of clinical chemistry parameters including: Lactate dehydrogenase.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 462 | 47
U/L
  End-of-stimulation visit: number analyzed (Participants) | 462 | 44
  End-of-stimulation visit | -13.6 (17.7) | -4.9 (17.0)
  End-of-cycle visit: number analyzed (Participants) | 457 | 47
  End-of-cycle visit | 1.2 (21.6) | -1.4 (14.8)

48. Secondary Outcome: Proportion of Subjects With Markedly Abnormal Changes of Clinical Chemistry Parameters: Phosphate, Potassium
Description: The table represents the percentage of participants in each group with normal baseline values and markedly abnormal end-of-stimulation or end-of-cycle visit values for phosphate and potassium.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 513 | 51
percentage of participants
  Phosphate (mmol/L) (End-of-stimulation visit): number analyzed (Participants) | 513 | 46
  Phosphate (mmol/L) (End-of-stimulation visit) | 0.2 | 0.0
  Potassium (mmol/L) (End-of-stimulation visit): number analyzed (Participants) | 504 | 47
  Potassium (mmol/L) (End-of-stimulation visit) | 0.2 | 0.0
  Phosphate (mmol/L) (End-of-cycle visit): number analyzed (Participants) | 504 | 50
  Phosphate (mmol/L) (End-of-cycle visit) | 0.2 | 0.0
  Potassium (mmol/L) (End-of-cycle visit): number analyzed (Participants) | 493 | 51
  Potassium (mmol/L) (End-of-cycle visit) | 1.0 | 0.0

49. Secondary Outcome: Changes in Haematology Parameters Compared to Baseline: Erythrocytes
Description: Blood samples were collected for the analysis of haematology parameter including: Erythrocytes.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 487 | 50
10^12 cells/L
  End-of-stimulation visit: number analyzed (Participants) | 480 | 42
  End-of-stimulation visit | -0.13 (0.22) | -0.04 (0.19)
  End-of-cycle visit | -0.18 (0.26) | -0.08 (0.22)

50. Secondary Outcome: Changes in Haematology Parameters Compared to Baseline: Leukocytes and Platelets
Description: Blood samples were collected for the analysis of haematology parameters including: Leukocytes and platelets.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 487 | 50
10^9 cells/L
  Leukocytes (End-of-stimulation visit): number analyzed (Participants) | 480 | 42
  Leukocytes (End-of-stimulation visit) | 1.203 (1.872) | -0.328 (1.521)
  Leukocytes (End-of-cycle visit) | 0.356 (2.106) | 0.154 (2.128)
  Platelets (End-of-stimulation visit): number analyzed (Participants) | 479 | 41
  Platelets (End-of-stimulation visit) | -7.2 (39.0) | -0.4 (43.7)
  Platelets (End-of-cycle visit): number analyzed (Participants) | 487 | 49
  Platelets (End-of-cycle visit) | 10.8 (48.7) | 0.9 (38.4)

51. Secondary Outcome: Changes in Haematology Parameters Compared to Baseline: Haemoglobin
Description: Blood samples were collected for the analysis of haematology parameters including: Haemoglobin.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 487 | 50
g/L
  End-of-stimulation visit: number analyzed (Participants) | 480 | 42
  End-of-stimulation visit | -3.44 (6.54) | -0.83 (5.83)
  End-of-cycle visit | -4.79 (8.11) | -1.98 (6.59)

52. Secondary Outcome: Changes in Haematology Parameters Compared to Baseline: Haematocrit
Description: Blood samples were collected for the analysis of haematology parameter including: Haematocrit.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 475 | 50
ratio
  End-of-stimulation visit: number analyzed (Participants) | 432 | 38
  End-of-stimulation visit | 0.0 (0.0) | 0.0 (0.0)
  End-of-cycle visit | 0.0 (0.0) | 0.0 (0.0)

53. Secondary Outcome: Changes in Haematology Parameters Compared to Baseline: Erythrocyte Mean Corpuscular Volume
Description: Blood samples were collected for the analysis of haematology parameter including: Erythrocyte mean corpuscular volume.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 475 | 50
femtoliters
  End-of-stimulation visit: number analyzed (Participants) | 432 | 38
  End-of-stimulation visit | 1.5 (3.1) | 1.3 (3.0)
  End-of-cycle visit | 1.1 (3.0) | 1.3 (3.1)

54. Secondary Outcome: Changes in Haematology Parameters Compared to Baseline: Erythrocyte Mean Corpuscular Hemoglobin
Description: Blood samples were collected for the analysis of haematology parameter including: Erythrocyte mean corpuscular hemoglobin.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: picogram
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 487 | 50
picogram
  End-of-stimulation visit: number analyzed (Participants) | 480 | 42
  End-of-stimulation visit | 0.1 (0.8) | 0.0 (0.7)
  End-of-cycle visit | 0.1 (0.9) | 0.0 (0.9)

55. Secondary Outcome: Changes in Haematology Parameters Compared to Baseline: Erythrocyte Mean Corpuscular Haemoglobin Concentration
Description: Blood samples were collected for the analysis of haematology parameter including: Erythrocyte mean corpuscular haemoglobin concentration.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 475 | 50
mmol/L
  End-of-stimulation visit: number analyzed (Participants) | 432 | 38
  End-of-stimulation visit | -0.3 (0.8) | -0.2 (0.7)
  End-of-cycle visit | -0.2 (0.8) | -0.2 (0.8)

56. Secondary Outcome: Changes in Haematology Parameters Compared to Baseline: Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/Leukocytes and Neutrophils/Leukocytes
Description: Blood samples were collected for the analysis of haematology parameters including: Basophils/leukocytes, eosinophils/leukocytes, lymphocytes/leukocytes, monocytes/leukocytes and neutrophils/leukocytes.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 487 | 50
percentage
  Basophils/leukocytes (End-of-stimulation visit): number analyzed (Participants) | 480 | 42
  Basophils/leukocytes (End-of-stimulation visit) | 0.01 (0.52) | 0.21 (0.54)
  Basophils/leukocytes (End-of-cycle visit) | 0.03 (0.45) | 0.07 (0.48)
  Eosinophils/leukocytes (End-of-stimulation visit): number analyzed (Participants) | 480 | 42
  Eosinophils/leukocytes (End-of-stimulation visit) | -0.52 (1.25) | -0.21 (1.19)
  Eosinophils/leukocytes (End-of-cycle visit) | -0.18 (1.29) | -0.15 (1.08)
  Lymphocytes/leukocytes (End-of-stimulation visit): number analyzed (Participants) | 480 | 42
  Lymphocytes/leukocytes (End-of-stimulation visit) | -6.25 (6.64) | 1.83 (5.13)
  Lymphocytes/leukocytes (End-of-cycle visit) | -1.86 (8.92) | -0.15 (6.59)
  Monocytes/leukocytes (End-of-stimulation visit): number analyzed (Participants) | 480 | 42
  Monocytes/leukocytes (End-of-stimulation visit) | -0.45 (1.74) | -0.35 (1.57)
  Monocytes/leukocytes (End-of-cycle visit) | 0.20 (1.65) | 0.06 (1.14)
  Neutrophils/leukocytes (End-of-stimulation visit): number analyzed (Participants) | 480 | 42
  Neutrophils/leukocytes (End-of-stimulation visit) | 7.22 (7.48) | -1.48 (5.49)
  Neutrophils/leukocytes (End-of-cycle visit) | 1.80 (9.88) | 0.18 (6.95)

57. Secondary Outcome: Proportion of Subjects With Markedly Abnormal Changes of Haematology Parameters: Leukocytes and Lymphocytes/Leukocytes.
Description: The table represents the percentage of participants in each group with normal baseline values and markedly abnormal end-of-stimulation or end-of-cycle visit values for Leukocytes and lymphocytes/leukocytes.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: From screening (baseline) to the end-of-stimulation visit and end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 477 | 49
percentage of participants
  Leukocytes (End-of-stimulation visit): number analyzed (Participants) | 447 | 39
  Leukocytes (End-of-stimulation visit) | 0.6 | 0.0
  Lymphocytes/leukocytes (End-of-stimulation visit): number analyzed (Participants) | 469 | 40
  Lymphocytes/leukocytes (End-of-stimulation visit) | 0.6 | 0.0
  Leukocytes (End-of-cycle visit): number analyzed (Participants) | 449 | 47
  Leukocytes (End-of-cycle visit) | 0.0 | 2.1
  Lymphocytes/leukocytes (End-of-cycle visit) | 0.4 | 2.0

58. Secondary Outcome: Frequency of Injection Site Reactions (Redness, Pain, Itching, Swelling and Bruising) Assessed by the Subject During the Stimulation Period
Description: Assessed by the participant during the stimulation period. Participants assessed the injection site reactions (redness, pain, itching, swelling and bruising) three times daily: immediately after the injection, 30 minutes after the injection and 24 hours after the injection.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: as for outcome 41
Measure: Number; unit: percentage of events
Units Other Than Participants: Total number of events
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
Number analyzed (Total number of events) | 63601 | 6545
percentage of events | 4.2 | 5.7

59. Secondary Outcome: Intensity of Injection Site Reactions (Redness, Pain, Itching, Swelling and Bruising) Assessed by the Subject During the Stimulation Period
Description: Assessed by the participant during the stimulation period as mild, moderate or severe.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: as for outcome 41
Measure: Number; unit: percentage of events
Units Other Than Participants: Total number of events
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
Number analyzed (Total number of events) | 63601 | 6545
percentage of events
  Mild injection site reaction | 4.1 | 5.7
  Moderate injection site reaction | 0.1 | 0.0458
  Severe injection site reaction | 0.0063 | 0

60. Secondary Outcome: Proportion of Subjects With Treatment-induced Anti-FSH Antibodies, Overall as Well as With Neutralizing Capacity
Description: Measured by presence of anti-FSH antibodies.
  95% Clopper-Pearson confidence interval has been reported in this endpoint.
Time Frame: Up to 28 days after end of the stimulation period
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants
  Treatment-induced anti-FSH antibodies (Overall) | 0.76 [0.21 to 1.94] | 0.00 [0.00 to 6.72]
  Treatment-induced anti-FSH antibodies with neutralizing capacity | 0 [NA to NA] — For participants with treatment-induced anti-FSH antibodies, none of the antibodies were of neutralizing capacity at any sampling time point. | 0 [NA to NA] — For participants with treatment-induced anti-FSH antibodies, none of the antibodies were of neutralizing capacity at any sampling time point.

61. Secondary Outcome: Frequency and Intensity of Immune-related AEs
Description: Standardised Medical Dictionary for Regulatory Activities (MedDRA) Queries (SMQs).
Time Frame: From time of signing informed consent until the end-of-cycle visit in the fresh cycle (approximately 6 months)
Population: as for outcome 41
Measure: Number; unit: events
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
events
  SMQ = Severe cutaneous adverse reactions | 3 | 0
  SMQ = Anaphylactic reaction | 5 | 0
  SMQ = Angioedema | 1 | 0
  SMQ = Hypersensitivity | 9 | 0
  Any general and local hypersensitivity reactions | 10 | 0

62. Secondary Outcome: Proportion of Subjects With Cycle Cancellations Due to an AE, Including Immune-related AEs, or Due to Technical Malfunctions of the Administration Pen
Description: For each participant the reason for cycle cancellation is recorded.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: Up to 20 stimulation days
Population: as for outcome 41
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants
  AE (including immune-related AEs) | 0 | 0
  Technical malfunctions of the administration pen | 0 | 0

63. Secondary Outcome: Proportion of Subjects With OHSS, Overall and by Grade, and Proportion of Subjects With Moderate/Severe OHSS
Description: Classification of grade was according to Golan's classification system, and all OHSS cases were graded as mild, moderate or severe.
  Data in this endpoint are presented for the fresh cycle.
Time Frame: ≤9 days after triggering of final follicular maturation (early OHSS), >9 days after triggering of final follicular maturation until 21-28 days after last IMP dose or up to ongoing pregnancy 8-9 weeks after transfer in pregnant participants (late OHSS)
Population: as for outcome 41
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants
  OHSS (any grade) | 3.8 | 0
  OHSS (moderate/severe) | 2.7 | 0

64. Secondary Outcome: Proportion of Subjects Hospitalized Due to OHSS and Proportion of Subjects Undergoing Paracentesis Due to OHSS
Description: Percentage of participants hospitalized or undergoing paracentesis due to OHSS are reported.
Time Frame: as for outcome 63
Population: as for outcome 41
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants
  Hospitalization | 0.2 | 0
  Paracentesis | 0.6 | 0

65. Secondary Outcome: Proportion of Participants With Multi-fetal Gestation in the Fresh Cycle
Description: Defined as pregnancy with more than one fetus. Among participants with ongoing pregnancy, percentage of participants with twin pregnancies are presented.
  '%' in the unit of measure refers to 'percentage'.
Time Frame: Up to 8-9 weeks after transfer
Population: as for outcome 1
Measure: Number; unit: % of participants with twin pregnancy
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 155
% of participants with twin pregnancy | 1.9

66. Secondary Outcome: Proportion of Cryopreserved Cycles With Multi-fetal Gestation
Description: Defined as pregnancy with more than one fetus. Among cryopreserved cycles with ongoing pregnancy, percentage of cycles with twin pregnancies are presented.
  '%' in the unit of measure refers to 'percentage'.
Time Frame: Up to 8-9 weeks after transfer
Population: as for outcome 1
Measure: Number; unit: % of cycles with twin pregnancy
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 184
% of cycles with twin pregnancy | 1.1

67. Secondary Outcome: Biochemical Pregnancy, Spontaneous Abortion, Ectopic Pregnancy (With and Without Medical/Surgical Intervention) and Vanishing Twins in the Fresh Cycle
Description: The percentage of participants with biochemical pregnancy, spontaneous abortion, ectopic pregnancy (with and without medical/surgical intervention) and vanishing twins in the fresh cycle are presented.
  The overall number of participants analyzed is the number of participants with positive βhCG.
  Data is not shown for placebo arm because no participants had a positive βhCG.
  '%' in the unit of measure refers to 'percentage'.
  Unit: Percentage of participants with early pregnancy loss.
Time Frame: Up to 8-9 weeks after transfer
Population: as for outcome 41
Measure: Number; unit: % of participants
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 184
% of participants
  Biochemical pregnancy | 9.2
  Spontaneous abortion | 6.5
  Induced abortion | 0.0
  Ectopic pregnancy | 0.0

68. Secondary Outcome: Biochemical Pregnancy, Spontaneous Abortion, Ectopic Pregnancy (With and Without Medical/Surgical Intervention) and Vanishing Twins in the Cryopreserved Cycles
Description: The percentage of cryopreserved cycles with biochemical pregnancy, spontaneous abortion, ectopic pregnancy (with and without medical/surgical intervention) and vanishing twins are presented.
  '%' in the unit of measure refers to 'percentage'.
  Data is not shown for placebo arm because no participants had a positive βhCG.
Time Frame: Up to 8-9 weeks after transfer
Population: as for outcome 41
Measure: Number; unit: % of cycles with early pregnancy loss
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 241
% of cycles with early pregnancy loss
  Biochemical pregnancy | 10.4
  Spontaneous abortion | 12.4
  Induced abortion | 0.0
  Ectopic pregnancy | 0.8

69. Secondary Outcome: Proportion of Participants With Technical Malfunctions of the Administration Pen
Description: Incidences of technical malfunctions of the administration pen were recorded.
Time Frame: Up to 20 stimulation days
Population: as for outcome 41
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
Number analyzed (Participants) | 525 | 53
percentage of participants | 0.2 | 0

ADVERSE EVENTS:
Time Frame: The AEs were recorded from time of signing informed consent to end-of-trial (up to Ongoing pregnancy visit (10-11 weeks after transfer)). Data for the AEs is presented for the fresh cycle and the cryopreserved cycle.
Description: Adverse events occurring after start of IMP and before the end-of-trial visit, or a pre-treatment AE or preexisting medical condition that worsens in intensity after start of FE 999049 or placebo treatment and before the end-of-trial visit (treatment-emergent AEs) are presented for the safety analysis set.
Arm/Group | FE 999049 (Follitropin Delta) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/525 | 0/53
Serious Adverse Events (participants affected / at risk) | 4/525 | 0/53
Other Adverse Events (participants affected / at risk) | 188/525 | 2/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | FE 999049 (Follitropin Delta) (N=525) | Placebo (N=53)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/278 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | FE 999049 (Follitropin Delta) (N=525) | Placebo (N=53)
Procedural pain (Injury, poisoning and procedural complications) | 150 (156) | 0 (0)
Morning sickness (Fresh cycle) (Pregnancy, puerperium and perinatal conditions) | 28 (34) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 30 (33) | 2 (2)
Morning Sickness (Cryopreserved cycle) (Pregnancy, puerperium and perinatal conditions) | 50/278 (60) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 31/278 (36) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 28/278 (30) | 0 (0)
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 22/278 (25) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT03740737/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT03740737/SAP_001.pdf